CLINICAL TRIAL: NCT03034564
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Droxidopa for Fatigue in Parkinson's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Site staffing
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-159
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Parkinson Disease; Fatigue; Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Fatigue; Parkinsonian Disorders | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Active group started 100 mg TID, increased by 100 mg per interval (i.e. 100 TID) every 2 days till on 600 TID, or until intolerable dose is achieved at which time the next highest dose will be maintained (increments of 100 TID will be used).
  Interventions: Drug: Northera
- 2 (Placebo Comparator): Dosing regimen identical to active group
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Northera
  Other Names: Droxidopa
  Arms: 1
Drug: Placebo Oral Tablet
  Arms: 2

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial comparing droxidopa to placebo for fatigue in Parkinson's Disease. The primary outcome measure is change in the Parkinson's Disease Fatigue Scale, a 16-item scale that measures the physical effects of fatigue as well as the impact of fatigue on daily functioning and activities, including socialization. Secondary outcomes are the PDQ-39, a 39-item self-report questionnaire assessing Parkinson's disease-specific health related quality over the last month in 8 different dimensions of function and well-being, and the Epworth Sleepiness Scale, a questionnaire querying 8 situations for which the subject will rate the likelihood of falling asleep. There will be a screening visit (SC), baseline visit (BL), 2 clinic visits at 6 and 12 weeks (V01, V02), and telephone contact at 4 weeks and 8 weeks (T1, T2). In-person visits will include review of informed consent, concomitant medication review, adverse event review, pill counts, vital signs (including supine blood pressure), and outcome measurements. Telephone visits will include review of informed consent, concomitant medication review, and adverse event review.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease
* Have normal kidney function (determined at screening visit by blood sample analysis), and no active medical diagnoses associated with fatigue
* No orthostatic symptoms (i.e. light headedness, blurred vision, and/or muscle weakness)
* No objective orthostasis (significant drop in blood pressure when standing)
* No supine hypertension (high blood pressure while laying down) judged to be of clinical significance by the investigator
* Well-controlled depression
* Stable dopaminergic medication regimen for 6 weeks prior to screening
* No concurrent use of fludrocortisone, midodrine, or other medications that may raise blood pressure
* PD Fatigue Scale Score of 50 or above

Exclusion Criteria:

* Diagnosis of Atypical Parkinsonism (having symptoms that mimic PD without a PD diagnosis)
* Prior Intolerance of droxidopa
* SNRI or TCA class (both antidepressant) medications (irrespective of indication)
* Use of activating agents (amantadine, modafinil, methylphenidate and related stimulants)
* Significant cardiac disease history
* Significant kidney disease history, or creatinine (a chemical found in the blood) greater than 1.5 mg/dl at baseline
* Poorly controlled depression
* Women who are pregnant or breastfeeding
* Significant history of Gastro Intestinal disease that may interfere with absorption (gastric bypass, inflammatory bowel disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01; Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease Fatigue Scale | Week 12
  16-item scale that measures the physical effects of fatigue as well as the impact of fatigue on daily functioning and activities, including socialization

SECONDARY OUTCOMES:
PDQ-39 | Week 12
  a 39-item self-report questionnaire assessing Parkinson's disease-specific health related quality over the last month in 8 different dimensions of function and well-being
Epworth Sleepiness Scale | Week 12
  a questionnaire querying 8 situations for which the subject will rate the likelihood of falling asleep

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGarry, MD, Principal Investigator — Cooper Health System
Locations (1):
- Cooper University Health System, Camden, New Jersey, United States